CLINICAL TRIAL: NCT03412409
Title: Reduced Intensity Conditioning Regimen for Elderly or High Comorbidity Burden Patients Receiving Haploidentical Hematopoietic Stem Cell Transplantation
Brief Title: RIC Regimen for Elderly or High Comorbidity Burden Patients Receiving Haplo-HSCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Director, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Haplo-RIC
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Acute Leukemia; Myelodysplastic Syndromes
Keywords: RIC regimen; comorbidity; elderly; haploidentical; transplant-related mortality
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Cytarabine; Busulfan; Cyclophosphamide; fludarabine; Semustine; Antilymphocyte Serum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RIC regimen (Experimental): Old patients or those have high comorbidity burden without identical sibling donor or unrelated donor would receive RIC haplo-HSCT.
  RIC preconditioning regimen consisted of cytarabine (2 g/m2/day, days -10 to -9), busulfan (3.2 mg/kg/day on days -8 to -6), cyclophosphamide (1.0 g/m2/day, days -5 to -4), fludarabine (30 mg/m-2/day, days -6 to -2), semustine (250 mg/m-2, day -3), and rabbit antithymocyte globulin (thymoglobulin, 2.5 mg/kg/d, days -5 to -2; Sanofi, France).
  Interventions: Drug: Cytarabine

INTERVENTIONS:
Drug: Cytarabine — RIC preconditioning regimen consisted of cytarabine (2 g/m2/day, days -10 to -9), busulfan (3.2 mg/kg/day on days -8 to -6), cyclophosphamide (1.0 g/m2/day, days -5 to -4), fludarabine (30 mg/m-2/day, days -6 to -2), semustine (250 mg/m-2, day -3), and rabbit antithymocyte globulin (thymoglobulin, 2.5 mg/kg/d, days -5 to -2; Sanofi, France).
  Other Names: Busulfan; Cyclophosphamide; Fludarabine; Semustine; Antithymocyte globulin

SUMMARY:
This study aimed to evaluate the efficacy of reduced intensity conditioning (RIC) regimen in elderly or high comorbidity burden patients who receive haploidentical hematopoietic stem cell transplantation (haplo-HSCT). Haplo-HSCT is an effective treatment option for patients who did not have identical sibling donor (ISD) or unrelated donor (URD). However, post-transplant transplant-related mortality (TRM) is one of the major causes for transplant failure, and the risk of TRM for old patients or those with high comorbidity burden was higher. RIC regimen may decrease the risk of TRM for haplo-HSCT recipients. The study hypothesis: Using RIC haplo-HSCT regimen in elderly patients or those with high comorbidity burden can reduce TRM and improve survival.

DETAILED DESCRIPTION:
RIC regimen was given for elderly patients or those with high comorbidity burden who would receive haplo-HSCT. The elderly patients were defined as older than 55 years. The burden of comorbidities in HSCT recipients was assessed based on the hematopoietic cell transplantation-specific comorbidity index (HCT-CI), and patients with score ≥3 were assigned as high burden. The primary end point was transplant-related mortality, and the secondary endpoints included overall survival, disease-free survival, relapse, engraftment, graft-versus-host disease (GVHD), and infections. Following time is 1 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 55 years or those with HCT-CI scores of ≥3, without ISD nor URD, receiving haplo-HSCT

Exclusion Criteria:

* patients having identical sibling or unrelated donors; patients with active infection; patients having organ failure; patients with poor compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Transplant-related mortality | Participants will be followed for an expected average of 1 years
  Death without disease progression or relapse

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, Principal Investigator — Institute of Hematology, Peking University
Locations (1):
- Peking University, Institute of Hematolgoy, Beijing, China

REFERENCES:
- [Derived] Sun W, Sun Y, Mo X, Ma R, He Y, Zhang Y, Chen Y, Wang F, Chen H, Chen Y, Yan C, Han W, Xu L, Wang Y, Zhang X, Liu K, Huang X. A novel and safe protocol for patients with severe comorbidity who undergo haploidentical hematopoietic stem cell transplantation: A single-center prospective study. J Transl Int Med. 2025 May 8;13(2):128-137. doi: 10.1515/jtim-2025-0018. eCollection 2025 Apr. PMID 40443407
- [Derived] Yu WJ, Sun YQ, Zhang XH, Xu LP, Mo XD, Lv M, Huang XJ, Wang Y. A novel reduced toxicity conditioning regimen for older myelodysplastic neoplasms patients undergoing haploidentical stem cell transplantation: a prospective cohort study. Am J Cancer Res. 2025 Jan 15;15(1):182-194. doi: 10.62347/OFXJ3130. eCollection 2025. PMID 39949947
- [Derived] Sun YQ, Han TT, Wang Y, Yan CH, Wang FR, Wang ZD, Kong J, Chen YH, Chen H, Han W, Chen Y, Zhang YY, Zhang XH, Xu LP, Liu KY, Huang XJ. Haploidentical Stem Cell Transplantation With a Novel Conditioning Regimen in Older Patients: A Prospective Single-Arm Phase 2 Study. Front Oncol. 2021 Feb 26;11:639502. doi: 10.3389/fonc.2021.639502. eCollection 2021. PMID 33718234